CLINICAL TRIAL: NCT03342677
Title: Evaluation of Gd-EOB-DTPA MRI for Detection and Characterization of Liver Nodules in Cirrhotic Patients Undergoing Liver Transplantation and Potential Impact on Transplant Eligibility
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN12-5803
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Cirrhosis; HCC; Primovist
MeSH Terms: conditions — Carcinoma, Hepatocellular; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): In this project, there is only one study group which comprises of patients with Hepatocellular Carcinoma (HCC) who will undergo Liver MRI with Primovist before hepatic transplantation.
  Interventions: Diagnostic Test: Primovist MRI

INTERVENTIONS:
Diagnostic Test: Primovist MRI — Utility of Gd-EOB-DTPA (Primovist) enhanced Liver MRI in HCC detection and characterization in cirrhotic patients will be studied.

SUMMARY:
Chronic liver disease including cirrhosis is one of the most important factors in the multi-step progression of hepatocarcinogenesis, from benign regenerative nodules to early hepatocellular carcinomas (HCCs) and finally to overt HCCs. Early diagnosis of HCC, differentiation from benign hepatocellular nodules, and surgical resection of the tumor or transplantation of the liver provide the best chance for long-term survival. Several studies have evaluated MRI enhanced with superparamagnetic iron oxide, gadolinium-based contrast material, or both, for the detection and differential diagnosis of focal hepatic lesions. However, the differentiation of HCC from benign and or borderline hepatocellular nodules remains difficult, particularly in patients with cirrhosis, because of the architectural distortion of liver parenchyma and the development of cirrhotic nodules, ranging from benign regenerative nodules to overt HCC, with overlapping imaging features. Recently, gadoxetic acid (gadoliniumethoxybezyl-diethylenetriamine pentaacetic acid; Primovist®, Bayer Health Care Pharmaceuticals), a gadolinium-based paramagnetic contrast agent that produces both dynamic and liver-specific hepatobiliary MRI studies has gained widespread use. Some studies have showed that gadoxetic acid-enhanced MRI allows the accurate detection and characterization of HCC. Investigators plan to assess this in particular as it is a question of great relevance. Execution of well conducted prospective studies will also clarify inclusion of Gd-EOB-DTPA enhanced MRI as the technique of choice in evaluation of patients at risk for HCC.

ELIGIBILITY:
Inclusion Criteria:

* a. Patients with liver cirrhosis enlisted for liver transplantation with high probability of undergoing transplantation within the ensuing 12 months

  b. Patients who are diagnosed or suspected with HCC and listed for liver transplant surgery with priority MELD (Model for End-Stage Liver Disease) points based on the cancer diagnosis, regardless of whether they have or have not received pre-transplant treatments (incl. RFA, TACE, and XRT)

  c. Subjects must be able to undergo MRI

Exclusion Criteria:

* a. GFR <30 mL/min/1.73 m2

  b. Elevated bilirubin (>3mg/dl)

  c. Pregnant and/or nursing women

  d. Contraindications to MRI such as pacemaker or ferromagnetic implants

  e. Hypersensitivity to Primovist or to any ingredient in the formulation or component of the container

  f. Younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-11-07 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of Gd-EOB-DTPA enhanced liver MRI and CT scan images in characterizing cirrhotic nodules and HCC in liver transplant candidates | 26 months

SECONDARY OUTCOMES:
Investigation of Gd-EOB-DTPA enhanced MRI efficacy in diagnosis and staging of HCC in cirrhotic patients and its potential impact on liver transplantation eligibility in patients who are liver transplant candidates | 26 months

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Jhaveri, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jhaveri KS, Babaei Jandaghi A, Bhayana R, Elbanna KY, Espin-Garcia O, Fischer SE, Ghanekar A, Sapisochin G. Prospective evaluation of Gadoxetate-enhanced magnetic resonance imaging and computed tomography for hepatocellular carcinoma detection and transplant eligibility assessment with explant histopathology correlation. Cancer Imaging. 2023 Feb 25;23(1):22. doi: 10.1186/s40644-023-00532-3. PMID 36841796